CLINICAL TRIAL: NCT03205449
Title: Parenting for Lifelong Health-Philippines: Randomized Controlled Trial of a Culturally-adapted Parenting Program on Reducing the Risk of Violence Against Children in Low-income Filipino Families With Children Aged 2 to 6 Years in Manila
Brief Title: Parenting for Lifelong Health (PLH) - Masayang Pamilya (MaPa) Evaluation Study
Acronym: PLH-MaPa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ateneo de Manila University (Other)
Collaborators: University of Oxford (Other); Philippine Ambulatory Pediatric Association (Unknown); Philippine Department of Social Welfare and Development (Unknown); Bangor University (Other); University of Cape Town (Other); International Child Protection Network (Other); The UBS Optimus Foundation (Unknown); UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AdMUREC_16_090
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Intervention Model Description: This study will use a randomised controlled trial design to test the effects of the Masayang Pamilya programme in comparison to participants allocated to a treatment as usual control group (N = 120 parents of children ages 2 to 6 years; 1:1 intervention to control group ratio).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MaPa Programme (Experimental): Masayang Pamilya Parenting Program: A 12-session, a group-based parenting programme focused on reducing violence against children and improving child wellbeing in low-income families with young children
  Interventions: Behavioral: Masayang Pamilya Para Sa Batang Pilipino Parenting Programme (MaPa)
- Treatment-as-usual (Active Comparator): Parenting Effectiveness Service programme: A family strengthening programme delivered by trained service providers on a monthly basis.
  Interventions: Other: Parenting Effectiveness Service

INTERVENTIONS:
Behavioral: Masayang Pamilya Para Sa Batang Pilipino Parenting Programme (MaPa) — The MaPa programme includes the following content: 1) spending one-on-one time with children; 2) describing actions and feelings for cognitive development and socio-emotional awareness; 3) using praise and rewards to encourage positive behaviour; 4) establishing limits through effective instruction giving and consistent household rules; 5) nonviolent discipline such as ignoring negative attention seeking behaviour, and consequences for noncompliance, rule-breaking, and aggressive behaviour; 6) problem solving with children; and 7) mindfulness based stress reduction for caregivers.
  Other Names: MaPa Programme
  Arms: MaPa Programme
Other: Parenting Effectiveness Service — Content uses a thematic manual that includes sessions on Filipino family dynamics, early childhood development, child behaviour management, marital relationships, prevention of child maltreatment, health care, nutrition, and government anti-poverty initiatives, as well as disaster preparedness. [12].
  Other Names: PES
  Arms: Treatment-as-usual

SUMMARY:
Parenting for Lifelong Health (PLH) Philippines Evaluation Study: Multisite randomised controlled trial to compare the efficacy of a culturally-adapted parenting programme, Masayang Pamilya, versus services as usual in the reduction of child maltreatment and improvement of child wellbeing in low-income Filipino families with children aged two to six years in Metro Manila (N = 120).

A previous study focused on adaptation and feasibility testing was conducted from January 2016 to February 2017. Community-based participatory approaches were used to culturally adapt the Sinovuyo programme to a Filipino context. A formative evaluation using qualitative in-depth interviews and focus group discussions with parents, as well as consultative workshops with service providers and other stakeholders, examined issues regarding the needs and concerns of Filipino parents, appropriateness of intervention components and delivery, and other specific cultural issues in order to balance "fidelity" to evidence-based practices with "fit" to the local context [11]. The Sinovuyo programme was then adapted into the MaPa programme with local materials and approaches developed to fit the Philippine cultural context based on findings from the formative evaluation.

DETAILED DESCRIPTION:
Over the past decade there have been increasing calls for the scale-up of evidence-based interventions in order to reduce the risk of violence against children in low- and middle-income countries (LMICs) [1]. In particular, parenting programmes for families with young children have been shown to be effective in reducing the risk of child maltreatment and improving child wellbeing with promising evidence emerging from low- and middle-income countries [2-4]. These group-based programmes typically aim to strengthen caregiver-child relationships through positive parenting and to help parents to manage child behaviour problems through effective, age-appropriate, nonviolent discipline strategies.

Despite the emerging evidence of the effectiveness of parenting interventions in reducing violence against children, many local governments and service providers in LMICs face multiple challenges implementing evidence-based parenting programs in resource poor contexts [5]. Parenting programmes are often too expensive to deliver effectively at scale in low-resource settings due to their complexity, intensity, and length [3]. Parenting programmes developed and evaluated in other contexts also may not fit the local service delivery context and may require adaptation to be relevant to the local culture of families. Additional programme content may also be necessary to address stress related to economic deprivation, high community violence, and parental distress. The process of delivery may also need to be simplified to improve participant engagement and the quality of delivery.

As a result, it is essential that programmes implemented in LMICs are 1) effective at reducing violence against children, 2) integrated within the existing service delivery system, 3) feasible and culturally acceptable to service providers and families, and 4) scalable in terms of their affordability, replicability, and sustainability while reaching a maximum number of beneficiaries. However, there are currently very few parenting programmes that meet these criteria in LMICs, such as the Philippines, where the need is the greatest [3].

The PLH Philippines Evaluation Study aims to fill this gap by examining the efficacy of a locally-adapted, evidence-based parenting programme, the Masayang Pamilya Para Sa Batang Pilipino Parenting Programme (MaPa), for families with children ages two to six years living in Metro Manila who are enrolled in the Philippine Department of Social Welfare and Development (DSWD) conditional cash transfer system.

Our overall objective is to use a randomised controlled trial design to test the efficacy of the MaPa programme in reducing the risk of child maltreatment while improving child socio-emotional development, child behaviour, and parental mental health in comparison to treatment as usual controls in Metro Manila.

Our primary objective is to examine the impact of the MaPa programme on the primary outcome of child maltreatment in comparison to treatment-as-usual controls at immediate post-intervention and at 1-year follow-up.

Our secondary objective is to examine the impact of the MaPa programme on proximal outcomes associated with increased risks of child maltreatment, namely, positive parenting, intrusive parenting, and harsh parenting in comparison to treatment-as-usual controls at immediate post-intervention and at 1-year follow-up.

Another secondary objective is to examine the impact of the MaPa programme at immediate post-intervention and at 1-year follow-up on child behaviour problems, child development outcomes (i.e., communication skills and socio-emotional development), parenting efficacy, parental wellbeing, parenting stress, parental depression, marital satisfaction, and intimate partner violence, in comparison to treatment as usual controls.

Our tertiary objective is to examine the implementation of the MaPa programme when delivered within the DSWD conditional cash transfer system in terms of programme adherence by parents (i.e., recruitment, enrolment, attendance, engagement, dropout, and completion) and delivery by service providers (i.e., competency and fidelity).

Our final objective is to examine predictors of programme adherence and associations between programme adherence and primary and secondary outcomes at immediate post-test and at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Primary caregiver responsible for the care of a child between the ages of two and six who is staying in the same household at least four nights a week in the previous month;
* Spend at least four nights a week in the same household as the child;
* Unemployed parent;
* Recipient of the 4Ps conditional cash transfer programme;
* Agreement to participate in the MaPa programme if allocated to the treatment condition;
* Provision of consent to participate in the full study.

Exclusion Criteria:

* Any adult who has already participated in the Parent Effectiveness Service;
* Any adult exhibiting severe mental health problems or acute mental disabilities;
* Any adult that has been referred to child protection services due to child abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Change in frequency of child maltreatment | Change from baseline at 7 months and at 19 months
  Child maltreatment will be measured using parent report of the ISPCAN Child Abuse Screening Tool-Intervention scale (19 items, ICAST-I), an adaptation of a multi-national and consensus-based survey instrument measuring parent-report the incidence and prevalence of child abuse and neglect (ICAST-P). It was validated in 6 LMIC and 7 languages (α = 0.77-0.88) and measures four types of abuse: physical, emotional and sexual abuse, as well as neglect. Response code for the ICAST-I was adapted to a scale from 0 to more than 8 times to assess the frequency of a certain behaviour in the past month. This study will assess incidence of child maltreatment by creating dichotomous variables for physical abuse, verbal abuse, and neglect, as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.

SECONDARY OUTCOMES:
Change in frequency of positive parenting | Change from baseline at 7 months and at 19 months
  Positive parenting behavior will be assessed using the Parenting of Young Children Scale (PARYC, 21 items) [5]. The PARYC measures the frequency of parent behavior over the previous month. Items are summed to create total frequency scores for positive parenting (7 items, e.g., "how often do you play with your child"), setting limits (7 items, e.g., "how often do you stick to your rules and not change your mind") and proactive parenting (7 items, e.g., "how often do you explain what you want your child to do in clear and simple ways"). It has been used with strong reliability in previous studies on the program adapted in this study [20].
Change in frequency of dysfunctional parenting | Change from baseline at 7 months and at 19 months
  Dysfunctional parenting behavior will be assessed using the Parenting Scale (PS, 30 items) [6]. This scale examines parent attitudes and beliefs regarding discipline practice. Responses are based on a 7-point Likert scale in which parents are presented with a situation and then are asked to choose between two alternative responses to a situation (1 = most effective; 7 = most ineffective; i.e., situation: "When I say my child can't do something;" response, score = 1: "I stick to what I said;" or response score = 7: "I let my child do it anyway"). Items are summed to create an overall score as well as for three subscales: Laxness, Over-reactivity, and Verbosity. The PS has been used widely to assess the effectiveness of parenting programs, including in low-resource settings such as Panama [21].
Change in levels of endorsement of physical punishment | Change from baseline at 7 months and at 19 months
  This study will ask one question from the UNICEF Multiple Indicator Cluster Survey [1] regarding parental attitudes to physical discipline based on a 5-point Likert scale of 0 to 4: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished." Caregivers will report whether they disagree or agree with the statement (0 = disagree strongly; 4 = agree strongly).
Change in number of daily child behavior problems and parenting behaviors | Change from baseline at 7 months and at 19 months
  An adapted version of Parent Daily Report Checklist (PDR, 44 items) will be used to assess day-to-day occurrences of child behavior problems and parenting behavior [12]. It was designed to avoid potential challenges parents may have in recalling events in retrospective scales, and has been used widely in multiple contexts as an assessment of child and parent behavior change during program delivery [46-49]. The PDR does not assess frequency of behavior but rather the occurrence (i.e., "Yes" or "No"). Parents indicate whether a child behavior occurred within the previous 24 hours (35 items, e.g., complaining, lying). In order to assess parenting behavior, this study will also ask parents about their own behavior (6 items, e.g., used physical discipline, or praised child) and self-efficacy (3 items, e.g., had a feeling that I could not cope with parenting).
Change in number of child behavior problems | Change from baseline at 7 months and at 19 months
  The Eyberg Child Behavior Inventory assesses child behavior problems [30]. This 36-item survey examines externalizing behavior problems in children ages 2 to 16 using both an Intensity Scale and Problem Scale. Parents are asked how often a specific behavior occurs and whether the behavior is considered a problem. Items based on the most typical child behavior problems. The Intensity Scale rates frequency of occurrence based on a 7-point Likert-like scale (1 = never occurs; 7 = always occurs). The Problem Scale measures whether the parent identifies a specific behavior as a problem (0 = no; 1 = yes). Both scales are summed up to create a total Intensity Score and Problem Score. The ECBI has been used extensively throughout the world as a diagnostic tool as well as to evaluate parenting programs in RCTs [31-34]. Clinical cut-off scores suggested for psychopathological problem behavior are 131 for the Intensity Score and 15 for the Problem Score [35].
Change in levels of child development - communication skills | Change from baseline at 7 months and at 19 months
  Child development will be assessed using the communication subscale of the parent-report version of the Ages and Stages Questionnaires, Version 3 (ASQ-3) [13]. This 6-item screening tool measures infant and toddler development of communication skills from 2 months to 6 years of age. Distinct items are administered according to the child's age in 2-month intervals rounded to the nearest interval. The ASQ-3 is administered via caregiver self-report based on "Yes," "Sometime," or "Not Yet" for each developmental milestone. In addition, if the caregiver is not sure of a specific item, s/he is given the opportunity to perform the task with his/her infant or toddler during the assessment. Items for each subscale are summed to create total scores as well as an overall indication of child development. Cut-off scores will be used based on international ASQ cut-offs according to the manual for normal development, borderline delay, and developmental delay [13].
Change in levels of child socio-emotional development | Change from baseline at 7 months and at 19 months
  Child socio-emotional development will be assessed using the parent-report version of the Ages and Stages Questionnaires: Social-Emotional, Version 2 (ASQ-SE2) [14, 36]. This screening tool was designed to specifically assess socio-emotional development for children from 1 month to 6 years of age. Questionnaires are administered to the parent depending on the age of the child (i.e., 24, 30, and 36 month intervals). Items examine seven domains of socio-emotional development: self-regulation, compliance, adaptive functioning, autonomy, affect, social-communication, and interaction with others. Parents report on whether the specific child behavior occurs "often or always," "sometimes," or "rarely or never," as well as whether the behavior is a concern for the parent (yes/no). The ASQ:SE has been used extensively as a global screening tool, including multiple low- and middle-income countries [37-41].
Change in levels of parent efficacy | Change from baseline at 7 months and at 19 months
  Parenting efficacy will be assessed using the Efficacy Subscale of the Parenting Sense of Competence Scale (8 items; PSOC-ES) [37]. The PSOC has been widely used in studies to evaluate parenting self-esteem, efficacy, or competence [37]. The PSOC Efficacy Subscale measures parental perception of competence, problem-solving ability, and capability in the parenting role (e.g., ""I honestly believe I have all the skills necessary to be a good mother/father to my child"). Each item is rated on a 6-point scale that ranges from 1 (strongly disagree) to 6 (strongly agree). Items are summed to create a total score of parental self-efficacy.
Change in levels of parenting stress | Change from baseline at 7 months and at 19 months
  Parenting stress will be measured using the Parenting Stress Index (PSI) (36 items) [8]. This scale has been used widely throughout the world [22-25], including prior use in low- and middle-income countries [26, 27]. Items include subscales for parental distress (e.g., "I often have the feeling that I cannot handle things very well"), parent-child dysfunction (e.g., "Sometimes I feel my child doesn't like me and doesn't want to be close to me"), and difficult child (e.g., "I feel that my child is very moody and easily upset"). Items are summed to create a total score for parenting stress as well as for each subscale.
Change in levels of parental depression | Change from baseline at 7 months and at 19 months
  The Depression, Anxiety, and Stress Scale (DASS) will assess caregiver depression. The DASS is a 21-item scale used as a screening tool to measure depression, anxiety, and stress in adults. Caregivers report on the frequency of depressive symptoms in the previous week using a Likert scale (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always; e.g., "I felt that I had nothing to look forward to"). Total DASS scores range from 0 to 63 with subscales from 0 to 21. Recommended cut-offs indicating severity of depression are 5-6 for mild, 7-10 for moderate, 11-13 for severe, and 14 and up for extremely severe. Cut-offs for anxiety are 4-5 for mild, 6-7 for moderate, 8-9 for severe, and 10 and up for extremely severe. Cut-offs for stress are 8-9 for mild, 10-12 for moderate, 13-16 for severe, and 17 and up for extremely severe.
Change in levels of parental wellbeing | Change from baseline at 7 months and at 19 months
  The WHO-5 Well-Being Scale (WHO-5) will measure parental psychological well-being [10]. This 5-item scale was derived using psychometric analyses from the longer 28-item WHO Well-Being Scale. The validation study of the WHO-5 showed 93% sensitivity and 64% specificity when compared with the General Health Questionnaire and the Patient Health Questionnaire [28]. Parents indicate the frequency that they experience well-being in the past month (e.g., "My daily life has been filled with things that interest me") based on a Likert scale from 0 to 5 ("At no time" to "All of the time"). Items are added up with scores ranging from 0 to 25.
Change in levels of parent dependency on alcohol | Change from baseline at 7 months and at 19 months
  Parental dependency on alcohol will be assessed by asking parents to report on alcohol consumption during the past month (1 item). Dependency is based on 3 or more drinks per day for female participants and 5 or more per day for male participants [48]. Due to the sensitive nature of these items, additional items dealing with other activities to reduce stress have been included in this section to encourage accuracy (3 items; e.g., "In the past month, have you been for a walk or done some other exercise to help you relax?").
Change in frequency of intimate partner violence | Change from baseline at 7 months and at 19 months
  Adult self-report of the victimhood of intimate partner violence will be assessed using an adapted version of the Revised Conflict Tactics Scale Short Form (CTS2S; 8 items) [42]. Items include the frequency of negotiation (e.g., "partner suggested compromise to an argument"), physical assault (e.g., "partner hit me with something"), and psychological aggression (e.g., "partner insulted or swore at me"). Answers are coded on a 5-point Likert scale of 0 to 4 (0 = never happened; 4 = more than 3 times in the past month). The CTS2S will determine an overall indication of IPV on a level of severity (sum of items) and prevalence (dichotomous variable indicating experience of conflict or not) as well as for each subscale.
Change in levels of marital satisfaction | Change from baseline at 7 months and at 19 months
  Adult report of marital satisfaction will be assessed using the Kansas Marital Satisfaction Scale (KMSS; 3 items) {Schumm, 1986 #3905}. The KMSS was developed as a validated but brief measurement of marital relations. Items include satisfaction with marriage, spouse or partner, and quality of the relationship with a spouse/partner. Responses options are coded on a 7-point Likert scale of 1 to 7 (1 = extremely dissatisfied; 7 = extremely satisfied). Total scores are created by summing the items. The KMSS has been found to correlate strongly with other measures relationship adjustment and quality of marriage, and showed strong internal reliability in the feasibility pilot of the MaPa programme (α = .89).
Change in levels of parent/child sleep | Change from baseline at 7 months and at 19 months
  Parent/child sleep will be assessed by asking parents to report average daily number of hours the parent and child slept in the previous five days. In order to increase the accuracy of self-report data, research assistants will ask the parent to report on the hours of sleep for each day including hours that the child sleeps during the day. Mean score for hours slept for both parent and child will be calculated summing each day and then dividing by the number of days (i.e., 5 days).

OTHER OUTCOMES:
Implementation fidelity | 7 months after baseline and at 19 months
  Implementation fidelity by program facilitators of the MaPa program will be measured using self-report checklists by program implementers will examine the extent to which core intervention components are delivered. These checklists will include specific activities for each session, such as home practice discussion and role-playing exercises. Then, in order to produce a basic level of fidelity, a ratio of program implementation to program design will be created for both self-report and observational scores [117]. According to Borrelli and colleagues, a standard of 80% program fidelity will be considered as "high treatment fidelity" [118].
Quality of delivery | 7 months after baseline and at 19 months
  Quality of delivery will be assessed using the Parenting for Lifelong Health Facilitator Assessment Tool (PLH-FAT) [60]. The PLH-FAT was developed by the study investigators and programme developers to assess the proficiency of programme delivery by facilitators as a prerequisite to certification. Seven standard behaviour categories are grouped into two scales based on the core activities (23 items) and process skills (28 items) as outlined in the programme manual [6]. Assessment of core activities includes quality of delivery during home activity review (14 items, e.g., "identify specific challenges when shared by at least one parent"), illustrated story discussion (7 items, e.g., "discuss possible solutions for negative stories"), and practicing skills (10 items, e.g., "debrief with the participants about experience and feelings"). Assessment of process skills includes modelling skills (6 items, e.g., "give positive, specific, and realistic instructions"), collaborative facilitation
Program adherence | 7 months after baseline and at 19 months
  Program adherence will be assessed by examining rates of enrolment, attendance, dropout, completion, and engagement of home activities. Enrolment rates will be based on the ratio of those allocated to the MaPa or PES intervention and those who attend at least one session. Mean attendance rates for enrolled participants will be determined based on the ratio of number of attended sessions to the total number of program sessions (MaPa = 12 sessions; PES = 9 sessions). Dropout rates for enrolled participants will be defined as the percentage of participants who fail to attend at least three consecutive sessions and do not attend any sessions at a later stage. Completion rates for the entire allocation group will be determined based on the number of enrolled participants who attend a cut-off threshold of at least 66% of the program. Engagement in home activities will be assessed using parent-report of home activity completion forms and by examining transcripts from parent group session.
Engagement in home activities | 7 months after baseline and at 19 months
  Engagement in home activities will be assessed using parent-report of home activity completion forms and by examining transcripts from parent group sessions. During each session, parents will report whether they were able to implement the assigned home activity activities from the previous week according to the intervention protocol. A weekly rate of engagement will be calculated based on the ratio of completed assignments to the number of parents in attendance during the session. Finally, an overall rating of engagement will be determined by summing each weekly rate. Although it is possible that non-attendees will also complete home activities, this study will only examine engagement based on those in attendance at any given session.
Participant satisfaction | 7 months after baseline and at 19 months
  Participant satisfaction will be examined for families who attend at least one session of the MaPa program [120]. Mean and standard deviation scores will be reported for the overall participation satisfaction scale (40 items), as well as for subscales (i.e., whether the program fulfilled their expectations, acceptability of delivery and teaching methods, acceptability of theoretical parenting techniques, and evaluation of program facilitators).
Program acceptability and participation | 7 months after baseline and at 19 months
  This study will also assess program acceptability and participation using qualitative in-depth interviews with intervention participants (n = 12) and focus groups with the facilitators (n = 8) in order to explore program acceptability. Participants will be purposively selected from the intervention group with the inclusion criteria of attending at least one intervention session. Selection will be based on those with high attendance (n = 3), those with low attendance (n = 3), those who dropout (n = 3), and those who do not enroll (n = 3). Interviews and focus groups will occur during the post-evaluation and examine the following themes: 1) participants observed change in parenting practices and child behavior at home during program; 2) acceptability and appropriateness of program materials, delivery, and key program components; and 3) existing barriers to participation during sessions and engagement in home practice and other activities.

CONTACTS AND LOCATIONS:
Overall Officials: Liane P Alampay, PhD, Principal Investigator — Ateneo de Manila University; Jamie M Lachman, PhD, Principal Investigator — University of Oxford; Cecilia Alinea, MD, Principal Investigator — Philippine Ambulatory Pediatric Association; Frances Gardner, PhD, Principal Investigator — University of Oxford; Judy Hutchings, PhD, Principal Investigator — Bangor University; Catherine Ward, PhD, Principal Investigator — University of Cape Town; Bernadette Madrid, MD, Principal Investigator — International Child Protection Network; Rosanne Jocson, PhD, Principal Investigator — Ateneo de Manila University
Locations (1):
- Barangay Western Bicutan, City of Taguig, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Anderson LS. Predictors of parenting stress in a diverse sample of parents of early adolescents in high-risk communities. Nurs Res. 2008 Sep-Oct;57(5):340-50. doi: 10.1097/01.NNR.0000313502.92227.87. PMID 18794718
- [Background] Armstrong R, Waters E, Moore L, Riggs E, Cuervo LG, Lumbiganon P, Hawe P. Improving the reporting of public health intervention research: advancing TREND and CONSORT. J Public Health (Oxf). 2008 Mar;30(1):103-9. doi: 10.1093/pubmed/fdm082. Epub 2008 Jan 19. PMID 18204086
- [Background] Baldwin SA, Murray DM, Shadish WR. Empirically supported treatments or type I errors? Problems with the analysis of data from group-administered treatments. J Consult Clin Psychol. 2005 Oct;73(5):924-35. doi: 10.1037/0022-006X.73.5.924. PMID 16287392
- [Background] Barlow J, Johnston I, Kendrick D, Polnay L, Stewart-Brown S. Individual and group-based parenting programmes for the treatment of physical child abuse and neglect. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD005463. doi: 10.1002/14651858.CD005463.pub2. PMID 16856097
- [Background] Bauer DJ, Sterba SK, Hallfors DD. Evaluating Group-Based Interventions When Control Participants Are Ungrouped. Multivariate Behav Res. 2008 Apr 2;43(2):210-236. doi: 10.1080/00273170802034810. PMID 20396621
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Borrelli B, Sepinwall D, Ernst D, Bellg AJ, Czajkowski S, Breger R, DeFrancesco C, Levesque C, Sharp DL, Ogedegbe G, Resnick B, Orwig D. A new tool to assess treatment fidelity and evaluation of treatment fidelity across 10 years of health behavior research. J Consult Clin Psychol. 2005 Oct;73(5):852-60. doi: 10.1037/0022-006X.73.5.852. PMID 16287385
- [Background] Castro FG, Barrera M Jr, Martinez CR Jr. The cultural adaptation of prevention interventions: resolving tensions between fidelity and fit. Prev Sci. 2004 Mar;5(1):41-5. doi: 10.1023/b:prev.0000013980.12412.cd. PMID 15058911
- [Background] Chen M, Chan KL. Effects of Parenting Programs on Child Maltreatment Prevention: A Meta-Analysis. Trauma Violence Abuse. 2016 Jan;17(1):88-104. doi: 10.1177/1524838014566718. Epub 2015 Jan 8. PMID 25573846
- [Background] Delgado-Rodriguez M, Llorca J. Bias. J Epidemiol Community Health. 2004 Aug;58(8):635-41. doi: 10.1136/jech.2003.008466. PMID 15252064
- [Background] Dunne MP, Zolotor AJ, Runyan DK, Andreva-Miller I, Choo WY, Dunne SK, Gerbaka B, Isaeva O, Jain D, Kasim MS, Macfarlane B, Mamyrova N, Ramirez C, Volkova E, Youssef R. ISPCAN Child Abuse Screening Tools Retrospective version (ICAST-R): Delphi study and field testing in seven countries. Child Abuse Negl. 2009 Nov;33(11):815-25. doi: 10.1016/j.chiabu.2009.09.005. Epub 2009 Oct 22. PMID 19853301
- [Background] Eames C, Daley D, Hutchings J, Whitaker CJ, Jones K, Hughes JC, Bywater T. Treatment fidelity as a predictor of behaviour change in parents attending group-based parent training. Child Care Health Dev. 2009 Sep;35(5):603-12. doi: 10.1111/j.1365-2214.2009.00975.x. Epub 2009 Jun 8. PMID 19508317
- [Background] Filgueiras A, Pires P, Maissonette S, Landeira-Fernandez J. Psychometric properties of the Brazilian-adapted version of the Ages and Stages Questionnaire in public child daycare centers. Early Hum Dev. 2013 Aug;89(8):561-76. doi: 10.1016/j.earlhumdev.2013.02.005. Epub 2013 Mar 16. PMID 23507472
- [Background] Garcia-Moreno C, Jansen HA, Ellsberg M, Heise L, Watts CH; WHO Multi-country Study on Women's Health and Domestic Violence against Women Study Team. Prevalence of intimate partner violence: findings from the WHO multi-country study on women's health and domestic violence. Lancet. 2006 Oct 7;368(9543):1260-9. doi: 10.1016/S0140-6736(06)69523-8. PMID 17027732
- [Background] Gardner F, Shaw DS, Dishion TJ, Burton J, Supplee L. Randomized prevention trial for early conduct problems: effects on proactive parenting and links to toddler disruptive behavior. J Fam Psychol. 2007 Sep;21(3):398-406. doi: 10.1037/0893-3200.21.3.398. PMID 17874925
- [Background] Gardner F, Hutchings J, Bywater T, Whitaker C. Who benefits and how does it work? Moderators and mediators of outcome in an effectiveness trial of a parenting intervention. J Clin Child Adolesc Psychol. 2010;39(4):568-80. doi: 10.1080/15374416.2010.486315. PMID 20589567
- [Background] Gardner MJ, Altman DG. Confidence intervals rather than P values: estimation rather than hypothesis testing. Br Med J (Clin Res Ed). 1986 Mar 15;292(6522):746-50. doi: 10.1136/bmj.292.6522.746. PMID 3082422
- [Background] Gershoff ET, Aber JL, Raver CC, Lennon MC. Income is not enough: incorporating material hardship into models of income associations with parenting and child development. Child Dev. 2007 Jan-Feb;78(1):70-95. doi: 10.1111/j.1467-8624.2007.00986.x. PMID 17328694
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Graham JW, Olchowski AE, Gilreath TD. How many imputations are really needed? Some practical clarifications of multiple imputation theory. Prev Sci. 2007 Sep;8(3):206-13. doi: 10.1007/s11121-007-0070-9. Epub 2007 Jun 5. PMID 17549635
- [Background] Henkel V, Mergl R, Kohnen R, Maier W, Moller HJ, Hegerl U. Identifying depression in primary care: a comparison of different methods in a prospective cohort study. BMJ. 2003 Jan 25;326(7382):200-1. doi: 10.1136/bmj.326.7382.200. No abstract available. PMID 12543837
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Heo KH, Squires J. Cultural adaptation of a parent completed social emotional screening instrument for young children: Ages And Stages Questionnaire-Social Emotional. Early Hum Dev. 2012 Mar;88(3):151-8. doi: 10.1016/j.earlhumdev.2011.07.019. Epub 2011 Sep 8. PMID 21855237
- [Background] Herth K. Hope as seen through the eyes of homeless children. J Adv Nurs. 1998 Nov;28(5):1053-62. doi: 10.1046/j.1365-2648.1998.00813.x. PMID 9840877
- [Background] Hinshaw SP. Intervention research, theoretical mechanisms, and causal processes related to externalizing behavior patterns. Dev Psychopathol. 2002 Fall;14(4):789-818. doi: 10.1017/s0954579402004078. PMID 12549704
- [Background] Hutchings J, Gardner F, Bywater T, Daley D, Whitaker C, Jones K, Eames C, Edwards RT. Parenting intervention in Sure Start services for children at risk of developing conduct disorder: pragmatic randomised controlled trial. BMJ. 2007 Mar 31;334(7595):678. doi: 10.1136/bmj.39126.620799.55. Epub 2007 Mar 9. PMID 17350966
- [Background] Kazdin AE, Holland L, Crowley M, Breton S. Barriers to Treatment Participation Scale: evaluation and validation in the context of child outpatient treatment. J Child Psychol Psychiatry. 1997 Nov;38(8):1051-62. doi: 10.1111/j.1469-7610.1997.tb01621.x. PMID 9413802
- [Background] Kerstjens JM, Bos AF, ten Vergert EM, de Meer G, Butcher PR, Reijneveld SA. Support for the global feasibility of the Ages and Stages Questionnaire as developmental screener. Early Hum Dev. 2009 Jul;85(7):443-7. doi: 10.1016/j.earlhumdev.2009.03.001. Epub 2009 Apr 7. PMID 19356866
- [Background] Kianifard F, Islam MZ. A guide to the design and analysis of small clinical studies. Pharm Stat. 2011 Jul-Aug;10(4):363-8. doi: 10.1002/pst.477. Epub 2010 Dec 8. PMID 21140524
- [Background] Knerr W, Gardner F, Cluver L. Improving positive parenting skills and reducing harsh and abusive parenting in low- and middle-income countries: a systematic review. Prev Sci. 2013 Aug;14(4):352-63. doi: 10.1007/s11121-012-0314-1. PMID 23315023
- [Background] Kraemer HC, Robinson TN. Are certain multicenter randomized clinical trial structures misleading clinical and policy decisions? Contemp Clin Trials. 2005 Oct;26(5):518-29. doi: 10.1016/j.cct.2005.05.002. PMID 15993653
- [Background] Kraemer HC, Wilson GT, Fairburn CG, Agras WS. Mediators and moderators of treatment effects in randomized clinical trials. Arch Gen Psychiatry. 2002 Oct;59(10):877-83. doi: 10.1001/archpsyc.59.10.877. PMID 12365874
- [Background] Labadarios D, Maunder E, Steyn N, MacIntyre U, Swart R, Gericke G, Nesamvuni E, Huskisson J, Vorster HH, Dannhauser A. National food consumption survey in children aged 1-9 years: South Africa 1999. Forum Nutr. 2003;56:106-9. No abstract available. PMID 15806819
- [Background] Lachman P, Poblete X, Ebigbo PO, Nyandiya-Bundy S, Bundy RP, Killian B, Doek J. Challenges facing child protection. Child Abuse Negl. 2002 Jun;26(6-7):587-617. doi: 10.1016/s0145-2134(02)00336-8. PMID 12201157
- [Background] Leung C, Sanders MR, Leung S, Mak R, Lau J. An outcome evaluation of the implementation of the Triple P-Positive Parenting Program in Hong Kong. Fam Process. 2003 Winter;42(4):531-44. doi: 10.1111/j.1545-5300.2003.00531.x. PMID 14979223
- [Background] Leung C, Leung S, Chan R, Tso K, Ip F. Child behaviour and parenting stress in Hong Kong families. Hong Kong Med J. 2005 Oct;11(5):373-80. PMID 16219957
- [Background] Lorenc T, Oliver K. Adverse effects of public health interventions: a conceptual framework. J Epidemiol Community Health. 2014 Mar;68(3):288-90. doi: 10.1136/jech-2013-203118. Epub 2013 Dec 13. PMID 24336237
- [Background] Martinez CR Jr, Eddy JM. Effects of culturally adapted parent management training on Latino youth behavioral health outcomes. J Consult Clin Psychol. 2005 Oct;73(5):841-51. doi: 10.1037/0022-006X.73.5.841. PMID 16287384
- [Background] McEachern AD, Dishion TJ, Weaver CM, Shaw DS, Wilson MN, Gardner F. Parenting Young Children (PARYC): Validation of a Self-Report Parenting Measure. J Child Fam Stud. 2012 Jun;21(3):498-511. doi: 10.1007/s10826-011-9503-y. PMID 22876108
- [Background] Mejia A, Calam R, Sanders MR. A pilot randomized controlled trial of a brief parenting intervention in low-resource settings in Panama. Prev Sci. 2015 Jul;16(5):707-17. doi: 10.1007/s11121-015-0551-1. PMID 25703382
- [Background] Mertens JR, Ward CL, Bresick GF, Broder T, Weisner CM. Effectiveness of nurse-practitioner-delivered brief motivational intervention for young adult alcohol and drug use in primary care in South Africa: a randomized clinical trial. Alcohol Alcohol. 2014 Jul-Aug;49(4):430-8. doi: 10.1093/alcalc/agu030. Epub 2014 Jun 4. PMID 24899076
- [Background] Mikton C, MacMillan H, Dua T, Betancourt TS. Integration of prevention of violence against children and early child development. Lancet Glob Health. 2014 Aug;2(8):e442-3. doi: 10.1016/S2214-109X(14)70233-5. Epub 2014 Jul 23. No abstract available. PMID 25103509
- [Background] Montgomery MR, Gragnolati M, Burke KA, Paredes E. Measuring living standards with proxy variables. Demography. 2000 May;37(2):155-74. PMID 10836174
- [Background] Morsbach SK, Prinz RJ. Understanding and improving the validity of self-report of parenting. Clin Child Fam Psychol Rev. 2006 Mar;9(1):1-21. doi: 10.1007/s10567-006-0001-5. PMID 16636897
- [Background] Pals SL, Murray DM, Alfano CM, Shadish WR, Hannan PJ, Baker WL. Individually randomized group treatment trials: a critical appraisal of frequently used design and analytic approaches. Am J Public Health. 2008 Aug;98(8):1418-24. doi: 10.2105/AJPH.2007.127027. Epub 2008 Jun 12. PMID 18556603
- [Background] Phillips AE, Gomez GB, Boily MC, Garnett GP. A systematic review and meta-analysis of quantitative interviewing tools to investigate self-reported HIV and STI associated behaviours in low- and middle-income countries. Int J Epidemiol. 2010 Dec;39(6):1541-55. doi: 10.1093/ije/dyq114. Epub 2010 Jul 14. PMID 20630991
- [Background] Potterton J, Stewart A, Cooper P. Parenting stress of caregivers of young children who are HIV Positive. Afr J Psychiatry (Johannesbg). 2007 Nov;10(4):210-4. doi: 10.4314/ajpsy.v10i4.30257. PMID 19588028
- [Background] Reid MJ, Webster-Stratton C, Beauchaine TP. Parent training in head start: a comparison of program response among African American, Asian American, Caucasian, and Hispanic mothers. Prev Sci. 2001 Dec;2(4):209-27. doi: 10.1023/a:1013618309070. PMID 11833925
- [Background] Runyan DK, Dunne MP, Zolotor AJ, Madrid B, Jain D, Gerbaka B, Menick DM, Andreva-Miller I, Kasim MS, Choo WY, Isaeva O, Macfarlane B, Ramirez C, Volkova E, Youssef RM. The development and piloting of the ISPCAN Child Abuse Screening Tool-Parent version (ICAST-P). Child Abuse Negl. 2009 Nov;33(11):826-32. doi: 10.1016/j.chiabu.2009.09.006. Epub 2009 Oct 24. PMID 19854511
- [Background] Bodenmann G, Cina A, Ledermann T, Sanders MR. The efficacy of the Triple P-Positive Parenting Program in improving parenting and child behavior: a comparison with two other treatment conditions. Behav Res Ther. 2008 Apr;46(4):411-27. doi: 10.1016/j.brat.2008.01.001. Epub 2008 Jan 5. PMID 18313033
- [Background] Straus MA, Douglas EM. A short form of the Revised Conflict Tactics Scales, and typologies for severity and mutuality. Violence Vict. 2004 Oct;19(5):507-20. doi: 10.1891/vivi.19.5.507.63686. PMID 15844722
- [Background] Streiner D, Geddes J. Intention to treat analysis in clinical trials when there are missing data. Evid Based Ment Health. 2001 Aug;4(3):70-1. doi: 10.1136/ebmh.4.3.70. No abstract available. PMID 12004740
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Vameghi R, Sajedi F, Kraskian Mojembari A, Habiollahi A, Lornezhad HR, Delavar B. Cross-Cultural Adaptation, Validation and Standardization of Ages and Stages Questionnaire (ASQ) in Iranian Children. Iran J Public Health. 2013 May 1;42(5):522-8. Print 2013. PMID 23802111
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Derived] Lachman JM, Alampay LP, Jocson RM, Alinea C, Madrid B, Ward C, Hutchings J, Mamauag BL, Garilao MAVFV, Gardner F. Effectiveness of a parenting programme to reduce violence in a cash transfer system in the Philippines: RCT with follow-up. Lancet Reg Health West Pac. 2021 Oct 5;17:100279. doi: 10.1016/j.lanwpc.2021.100279. eCollection 2021 Dec. PMID 34734199